

# +AGIL Barcelona: Integrated Care for Frail Older Adults Living in the Community

### **Participant Consent**

I declare that I have been invited to participate in the research study: "+AGIL Barcelona: Integrated Care for Frail Older Adults Living in the Community," conducted in the Larrard, Vila Olímpica, and Barceloneta Primary Care Centers. This study is made possible by the coordination of professionals from these centers and Parc Sanitari Pere Virgili.

Before signing this consent, I was informed that this study will evaluate the results and benefits of a multidimensional intervention, including lifestyle changes, medication adjustments, and strategies aimed at improving health and physical capacity.

The study is conducted in the aforementioned primary care centers. The researchers will perform an initial evaluation, followed by follow-up visits at 3 and 6 months from the first visit. Researchers may also contact me for individual or group interviews, which may be recorded with my explicit consent. If I agree to the recording, the images will be used solely for the purposes of this project.

I was also informed that participation is voluntary and anonymous and that I will not receive any financial compensation. Although I participate freely and voluntarily, I understand that I may withdraw from the study at any time without consequences.

Withdrawal from the study can be done at any point by verbally notifying the study researchers. If I decide to withdraw voluntarily, I may request that my data, both in paper and electronic formats, be traced and completely deleted.

The study data, particularly those relating to my personal and medical history, will remain confidential and will only be used for this research. My data will be stored in the file "Patient File of Parc Sanitari Pere Virgili," approved by decree of the Generalitat de Catalunya (DOGC CVE-DOGC-A-14038026-2014), with file number 204200205-H. The file complies with the guarantees provided under the Spanish Data Protection Law (LOPDP



15/1999). I understand that my data will be processed in accordance with the Data Protection Act (15/1999) and the Basic Law on Patient Autonomy and Rights and Obligations in Information and Clinical Documentation (41/2002).

Thus, I give my consent to participate in the study and declare that I have been informed, have read this consent, have had the opportunity to ask questions, and have received satisfactory answers to my questions.

| In Barcelona, on of | , 2022 |
|--------------------------|--------|
| Participant's ID: | |
| | - |
| Informant's ID: | _ |
| Participant's Signature: | |
| Informant's Signature: | |



# +AGIL Barcelona: Integrated Care for Frail Older Adults Living in the Community - ARCO Form

In accordance with Organic Law 15/1999, of December 13, on the Protection of Personal Data, and related regulations, we inform you that the personal data collected in this study will be included in a personal data file managed by Parc Sanitari Pere Virgili, with the sole purpose of conducting the mentioned clinical trial. If you wish to exercise your rights of access, rectification, or cancellation in the future, please complete this form and submit it to any of the researchers responsible for the study.

#### FILE MANAGER INFORMATION:

Parc Sanitari Pere Virgili

Carrer d'Esteve Terradas, 30, Parc Sanitari Pere Virgili, Tramuntana Building, 2nd floor,

I, \_\_\_\_\_, of legal age, residing at \_\_\_\_\_, in the city of

08023 Barcelona

Tax ID: S0800012G

(Dr. José Arturo Míguez Rey, Manager)

#### DATA OF THE INTERESTED PARTY OR LEGAL REPRESENTATIVE

| , province of, postal code, with ID/NIL |
|---|
| (copy attached), hereby exercise my data protection rights regarding the |
| data collected as part of the study "Integrated Primary and Geriatric Care with |
| Longitudinal Vision: +ÁGIL Barcelona, a Pragmatic Clinical Trial," in accordance with |
| Organic Law 15/1999. |
| I REQUEST (check the applicable options): |
| • Access to my data within one month from the receipt of this request, and |
| provision of information related to my participation in the study. |
| ullet Rectification of personal data within ten days from the receipt of this |
| request, with written notification of the corrections made. |



| Signat | ture: |
|---|---|
| In | , on, 2022. |
| • | Opposition to the inclusion of my personal data in the mentioned file within ten days from the receipt of this request, with written notification of the results. |
| | request, with written notification of the deletion. |
| • | $\square$ Cancellation of personal data within ten days from the receipt of this |